CLINICAL TRIAL: NCT00806364
Title: Normal Blood, Bone Marrow and Buccal Mucosa Protocol
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090049; 09-I-0049
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-11

CONDITIONS: Non-atopic; Atopic; Healthy; Normal; Allergy
Keywords: Skin; HV; Allergy; Healthy Volunteer; Non-atopic
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, stool, buccal/nasal/skin swabs, saliva, and tissue

GROUPS / COHORTS (1):
- 1: Blood, skin, stool/rectal swabs, buccal mucosa and bone marrow aspirate samples from approximately 250 healthy volunteer donors

SUMMARY:
This protocol is designed to provide blood, buccal mucosa and bone marrow aspirate samples from approximately 250, healthy volunteer donors for use in in vitro studies of mast cells, mastocytosis, and allergic diseases. Non-atopic donors will be recruited to donate blood, bone marrow, and/or buccal mucosa samples using conventional techniques. The investigational nature of the studies in which their blood, bone marrow and buccal mucosa samples will be used, as well as the risks and benefits of the donation process will be explained to all donors, and a signed informed consent document will be obtained. Donors will be compensated according to an established schedule based on the duration and discomfort of the donations. Samples provided through this protocol will be used solely for in vitro research. Blood, bone marrow, and buccal mucosa samples will be assigned a unique product number and the study investigators listed on this protocol will serve as the custodians of the code that links the product with a donor s identity. The nature of the in vitro studies in which the blood collected in this study will be used is not the subject of this protocol and will be described in general terms only. The samples will be used in several Institutional Review Board (IRB)-approved Laboratory of Allergic Diseases (LAD) protocols. This protocol is designed to assure adequate and complete informed consent, counseling, and protection of the study subjects according to IRB, Office of Human Subjects Research (OHSR), Office for Human Research Protections (OHRP) and other applicable Federal regulatory standards.

DETAILED DESCRIPTION:
This protocol is designed to provide blood, skin, stool/rectal swabs, buccal mucosa and bone marrow aspirate samples from approximately 250 healthy volunteer donors for use in in vitro studies such as studies of cells of the immune system, mastocytosis, and allergic diseases. Participants will donate samples using conventional techniques. The investigational nature of the studies in which samples will be used, as well as the risks and benefits of the donation process, will be explained to all donors, and a signed informed consent document will be obtained. Donors will be compensated according to an established schedule based on the duration and discomfort of the donations. Samples provided through this protocol will be used solely for in vitro research. Samples will be assigned a unique product number, and the study investigators will serve as the custodians of the code that links the product with a donor s identity. The nature of the in vitro studies in which the blood collected in this study will be used is not the subject of this protocol and will be described in general terms only. The samples will be used in several Institutional Review Board (IRB)-approved Laboratory of Allergic Diseases (LAD) protocols. This protocol is designed to assure adequate and complete informed consent, counseling, and protection of the study subjects according to IRB, Office of Human Subjects Research Protections, Office for Human Research Protections (OHRP) and other applicable Federal regulatory standards.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Ability to sign informed consent.

Healthy male or female between 18-65 years of age.

Willing to have samples stored for future research.

PARTICIPANT EXCLUSION CRITERIA:

History of an immune deficiency, such as HIV infection or cancer.

History of chronic hepatitis B and/or C infection.

History of chronic anemia.

A known clotting disorder or taking medications that interfere with blood clotting, such as: aspirin, heparin, or Coumadin*

Current pregnancy.

Have taken an investigational drug in the last 6 months that may affect the normal process of blood cells.

Any condition that in the view of the principal investigator (PI) would make the subject unsuitable for enrollment in this study.

* Coumadin and/or heparin treatment will not be stopped so that a subject can participate in this protocol. If Coumadin or heparin was recently discontinued, a subject can be enrolled, but no bone marrow procedures will be performed until the PT and the PTT are within normal range. For other agents that interfere with blood clotting without prolonging the PT, a 7-day washout period will be required before bone marrow sampling.

BONE MARROW PROCEDURE EXCLUSION CRITERIA

hemoglobin less than the NIH Clinical Center Clinical Research Information System (CRIS) normal range.

Platelets less than 100,000/mm(3).

PT or PTT greater than the NIH Clinical Center CRIS normal range

Positive b-HCG.

EKG changes suggestive of cardiovascular disease.

unable or unwilling to have bone marrow biopsy performed without use of conscious sedation, and use of only local anesthetic during procedure

Any other lab value which may put the subject at risk during the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2009-03-26 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
To provide an Institutional Review Board (IRB)-approved mechanism for the collection of peripheral blood, skin, bone marrow and/or buccal mucosa samples from healthy volunteer donors for use in in vitro studies. | 12/31/2030
  To provide an Institutional Review Board (IRB)-approved mechanism for the collection of peripheral blood, skin, bone marrow and/or buccal mucosa samples from healthy volunteer donors for use in in vitro studies.

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh D Komarow, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Vidal C, Gude F, Boquete O, Fernandez-Merino MC, Meijide LM, Rey J, Lojo S, Gonzalez-Quintela A. Evaluation of the phadiatop test in the diagnosis of allergic sensitization in a general adult population. J Investig Allergol Clin Immunol. 2005;15(2):124-30. PMID 16047713
- [Background] Hamilton RG, Adkinson NF Jr. 23. Clinical laboratory assessment of IgE-dependent hypersensitivity. J Allergy Clin Immunol. 2003 Feb;111(2 Suppl):S687-701. doi: 10.1067/mai.2003.123. PMID 12592314
- [Background] Standards for blood banks and transfusion services. QRB Qual Rev Bull. 1977 Dec;3(12):17,22. No abstract available. PMID 414187
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0049.html